CLINICAL TRIAL: NCT03856216
Title: Addition of Inotuzumab Ozogamicin Pre- and Post-Allogeneic Transplantation
Brief Title: Inotuzumab Ozogamicin and Chemotherapy in Treating Patients With Leukemia or Lymphoma Undergoing Stem Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: <75% participation
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0860; NCI-2019-00531 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0860 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-02-21; First posted 2019-02-27 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Acute Lymphoblastic Leukemia; B Acute Lymphoblastic Leukemia; Lymphocytic Neoplasm; Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma | interventions — Bone Marrow Transplantation; Bendamustine Hydrochloride; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine; Inotuzumab Ozogamicin; Melphalan; Peripheral Blood Stem Cell Transplantation; Rituximab; CT-P10; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (inotuzumab ozogamicin, chemotherapy, transplant) (Experimental): Recipients of haploidentical or mismatched unrelated stem cell transplant: Patients will receive inotuzumab ozogamicin intravenously (IV) over 1 hour on day -13, fludarabine IV over 1 hour on days -5 to -2, melphalan IV over 30 minutes on day -3 to -2, total body irradiation on day -1, and tacrolimus IV continuously beginning on day -2 then orally (PO) once daily (QD) or twice daily (BID) for about 6 months. Patients also receive bone marrow or peripheral blood progenitor cells IV on day 0. Patients receive cylophosphamide IV over 3 hours and mesna IV on days +3 to +4 and filgrastim-sndz subcutaneously (SC) QD beginning 1 week after the transplant until blood cell levels return to normal.
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Biological: Filgrastim-sndz; Drug: Fludarabine; Biological: Inotuzumab Ozogamicin; Drug: Melphalan; Procedure: Peripheral Blood Stem Cell Transplantation; Biological: Rituximab; Drug: Tacrolimus
- Group II (inotuzumab ozogamicin, chemotherapy, transplant) (Experimental): Recipients of haploidentical or mismatched unrelated stem cell transplant: Patients will receive inotuzumab ozogamicin intravenously (IV) over 1 hour on day -13, fludarabine IV over 1 hour on days -5 to -2, melphalan IV over 30 minutes on day -3 to -2, total body irradiation on day -1, and tacrolimus IV continuously beginning on day -2 then orally (PO) once daily (QD) or twice daily (BID) for about 6 months. Patients also receive bone marrow or peripheral blood progenitor cells IV on day 0. Patients receive cylophosphamide IV over 3 hours and mesna IV on days +3 to +4 and filgrastim-sndz subcutaneously (SC) QD beginning 1 week after the transplant until blood cell levels return to normal.
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Drug: Bendamustine; Biological: Filgrastim-sndz; Drug: Fludarabine; Biological: Inotuzumab Ozogamicin; Procedure: Peripheral Blood Stem Cell Transplantation; Biological: Rituximab; Drug: Tacrolimus

INTERVENTIONS:
Procedure: Allogeneic Bone Marrow Transplantation — Given IV
  Other Names: Allo BMT; Allogeneic Blood and Marrow Transplantation; Allogeneic BMT
Drug: Bendamustine — Given IV
  Other Names: SDX-105
  Arms: Group II (inotuzumab ozogamicin, chemotherapy, transplant)
Biological: Filgrastim-sndz — Given IV
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Zarxio
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Biological: Inotuzumab Ozogamicin — Given IV
  Other Names: Besponsa; CMC-544; Way 207294; WAY-207294
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
  Arms: Group I (inotuzumab ozogamicin, chemotherapy, transplant)
Procedure: Peripheral Blood Stem Cell Transplantation — Given IV
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Drug: Tacrolimus — Given IV and PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic

SUMMARY:
The goal of this phase II clinical study is to learn about the safety of inotuzumab ozogamicin when given with fludarabine, with or without bendamustine, melphalan, and rituximab before and after a stem cell transplant. Researchers also want to learn if inotuzumab ozogamicin when given after a stem cell transplant can help control leukemia and lymphoma. Inotuzumab ozogamicin is a monoclonal antibody, called inotuzumab, linked to a chemotherapy drug called ozogamicin. Inotuzumab attaches to CD22-positive cancer cells in a targeted way and delivers ozogamicin to kill them. Giving chemotherapy before a bone marrow or peripheral blood stem cell transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. Sometimes the transplanted cells from a donor attack the body's normal cells (called graft-versus-host disease). Giving tacrolimus and filgrastim before or after the transplant may stop this from happening. Fludarabine, bendamustine, melphalan, and rituximab are commonly given before stem cell transplants. Giving inotuzumab ozogamicin with chemotherapy may work better in treating patients with leukemia or lymphoma undergoing stem cell transplantation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety of the addition of inotuzumab ozogamicin (IO) pre- and post-allogeneic transplantation in patients with CD22-positive hematological malignancies.

SECONDARY OBJECTIVES:

I. Overall survival, progression-free survival and relapse rates. II. Treatment-related mortality. III. Cumulative incidence of acute and chronic graft-versus-host disease (GVHD).

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP I: Patients with acute lymphoblastic leukemia (ALL) and aggressive lymphoma receive inotuzumab ozogamicin intravenously (IV) over 1 hour on day -13, fludarabine IV over 1 hour on days -5 to -2, melphalan IV over 30 minutes on day -2, and tacrolimus IV continuously beginning on day -2 then orally (PO) once daily (QD) or twice daily (BID) for about 6 months. Patients also receive bone marrow or peripheral blood progenitor cells IV on day 0. Patients receive cylophosphamide IV over 3 hours and mesna IV on days +3 to +4 and filgrastim-sndz subcutaneously (SC) QD beginning 1 week after the transplant until blood cell levels return to normal.

GROUP II: Patients with indolent lymphoma receive inotuzumab ozogamicin IV over 1 hour on day -13, fludarabine IV over 1 hour and bendamustine IV over 30 minutes to 1 hour on days -5 to -3, and tacrolimus IV continuously beginning on day -2 then PO QD or BID for about 6 months. Patients also receive bone marrow or peripheral blood progenitor cells IV on day 0. Patients then receive rituximab IV over 4-6 hours on days 1 and 8, cyclophosphamide IC over 3 hours and mesna IV on days +3 to +4, and filgrastim-sndz SC once a day beginning 1 week after the transplant.

MAINTENANCE: Between 45 and 100 days after stem cell transplantation, all patients receive inotuzumab ozogamicin IV over 1 hour on days 1 and 2. Beginning 28 to 100 days after start of first cycle, patients receive inotuzumab ozogamicin IV over 1 hour on days 1 and 2 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

GROUP III: Recipients of haploidentical or mismatched unrelated stem cell transplant: Patients will receive inotuzumab ozogamicin intravenously (IV) over 1 hour on day -13, fludarabine IV over 1 hour on days -5 to -2, melphalan IV over 30 minutes on day -3 to -2, total body irradiation on day -1, and tacrolimus IV continuously beginning on day -2 then orally (PO) once daily (QD) or twice daily (BID) for about 6 months. Patients also receive bone marrow or peripheral blood progenitor cells IV on day 0. Patients receive cylophosphamide IV over 3 hours and mesna IV on days +3 to +4 and filgrastim-sndz subcutaneously (SC) QD beginning 1 week after the transplant until blood cell levels return to normal.

ELIGIBILITY:
Inclusion Criteria:

* Participants age 12 to 75.
* English and non-English speaking participants are eligible.
* CD22+ lymphoid malignancies including B-ALL
* Eligible to receive a reduced-intensity alloSCT

Participants with:

* Indolent lymphoma participants who failed conventional treatment; or,
* Acute lymphoblastic leukemia (ALL), aggressive lymphoma, indolent lymphoma in transformation, or those who have failed ≥ three small molecule inhibitors
* Donor: HLA compatible (8/8 match) related or matched unrelated donor (HLA-A, B, C, DRB1) or mismatched MUD (7/8 match) or haploidentical
* Performance status of 0 to 2, Lansky ≥ 80 for < 16 years and Karnofsky ≥ 80 for ≥ 16 years of age.
* Adequate organ function at time of study entry

  1. Creatinine less than or equal to 1.6 mg/dL
  2. Bilirubin less than 1.6 mg/dL
  3. SGPT < 2 x UL
  4. Ejection fraction >/= 40%
  5. FEV1, FVC and cDLCO >/= 40%
* Negative Beta HCG test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization) or currently breast-feeding. Pregnancy testing is not required for post-menopausal or surgically sterilized women.

Exclusion Criteria:

* Human immunodeficiency virus (HIV) positive.
* Prior autologous transplant less than 1 year prior to consent.
* Active and uncontrolled disease/infection.
* Unable or unwilling to sign consent.
* Current active hepatic or biliary disease (with exception of Gilbert's syndrome).
* Active hepatitis B or C.
* Recent systemic chemotherapy or radiation within 3 weeks of study entry (intrathecal therapy is allowed).

Standard biological agents such as rituximab, TKIs such as ibrutinib and venetoclax are allowed to be given within 3 days prior to receiving inotuzumab ozogamicin. Blinatumomab is allowed to be given until 1 week prior to Day -13 inotuzumab ozogamicin on study.

* Prior inotuzumab ozogamicin within 3 weeks of study entry.
* Peripheral blast count of greater than 10 K/mL.
* QTcF interval > 470 ms.
* Participants with cognitive impairments and/or any serious unstable pre-existing medical condition or psychiatric disorder that can interfere with safety or with obtaining informed consent or compliance with study procedures.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Incidence of grade 3 or higher renal, hepatic, cardiac, pulmonary, or neurologic toxicity | Up to 30 days after cycle 1 of maintenance therapy
  Will be assessed using the Bayesian method of Thall, Simon, and Estey. At the end of the trial, the rates of severe toxicity will be summarized, and analyses will be performed to assess the relationship between each toxicity endpoint and covariates of interest using logistic regression.

SECONDARY OUTCOMES:
Treatment-related mortality (TRM) | Up to 2 years
  The cumulative incidence of TRM will be assessed in a competing risks framework with the competing risk of disease relapse. Regression models will be fit to assess the relationship between each and covariates of interest using the method of Fine and Gray.
Relapse | Up to 2 years
Overall survival (OS) | Up to 2 years
  The distribution of OS will be assessed using the Kaplan-Meier method, and distributions will be compared using the log-rank test. Cox proportional hazards regression models will be fit to assess the relationship between OS and covariates of interest.
Progression-free survival (PFS) | Up to 2 years
  The distribution of PFS will be assessed using the Kaplan-Meier method, and distributions will be compared using the log-rank test. Cox proportional hazards regression models will be fit to assess the relationship between PFS and covariates of interest.
Acute graft versus host disease (GVHD) | Up to 2 years
  The cumulative incidence of acute GvHD will be assessed in a competing risks framework with competing risks of death without relapse and disease relapse. The method of Fine and Gray will be used to assess the association between GvHD and covariates of interest.
Chronic GVHD | Up to 2 years
  The cumulative incidence of chronic GvHD will be assessed in a competing risks framework with competing risks of death without relapse and disease relapse. The method of Fine and Gray will be used to assess the association between GvHD and covariates of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Issa F Khouri, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2025-06-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT03856216/ICF_001.pdf